CLINICAL TRIAL: NCT00000325
Title: Psychostimulant Abuse - Novel Treatment Approaches
Brief Title: Psychostimulant Abuse - Novel Treatment Approaches - 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Mclean Hospital (Other)
Purpose: Treatment
Other Study IDs: NIDA-10757-1; R01-10757-1
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2002-12

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Gonadotropin-Releasing Hormone

INTERVENTIONS:
Behavioral: Gonadorelin

SUMMARY:
To determine if acute assessments of profasi and factrel affect plasma cocaine levels and cocaine-induced behavioral changes in men.

ELIGIBILITY:
Please contact site for information.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0
Dates: Study Completion 2001-12

CONTACTS AND LOCATIONS:
Overall Officials: Jack Mendelson, M.D., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Dept. of Psychiatry, Belmont, Massachusetts, United States